CLINICAL TRIAL: NCT03026595
Title: The Profile of the Depression and it's Intervention Strategy in Patients With Parkinson's Disease in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-16-047
Record Dates: First submitted 2017-01-11; First posted 2017-01-20 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Depression is considered to be the most common neuropsychiatric disturbance of PD. In this study, investigators will summarize the treatment profile of PD depression to see if PD depression is properly treated according to guideline.

DETAILED DESCRIPTION:
Depression is considered to be the most common neuropsychiatric disturbance of PD. Prevalence rates of depressive disorders in Parkinson's disease(PD) vary widely across studies, ranging from 2.7% to more than 90%. A systematic review of the 36 articles concerning PD and depression indicates that the weighted frequency of depressive PD was 52%.

Investigators' previous study on non-motor symptoms in 81 Chinese PD patients demonstrated that prevalence of loss of interest and depression(sadness) were 48.7% and 36.7% by Non-motor symptoms questionnaire (NMSQuest) separately, which was similar to average global data. But another Chinese data published in 2008 showed that the prevalence of depression in PD patients was only 12%, no statistical difference with controls(2%). Thus, investigators plan to initiate a larger study to understand if PD depression in China is similar to it in western countries.

Depression would occur at the early stage of the disease or proceed the motor symptoms, usually accompanied with other non-motor symptoms including apathy, sleep disorder, cognitive impairment, and etc. The effects of depression on quality of life might refer to a wider range. There is lack of solid data to reveal the harm of depression on quality of life of PD patients and caregivers. In clinical practice, the disease burden of PD depression is usually underestimated by physicians and patients.

Although PD depression affects QoL of patients and caregivers, PD depression would be relieved by medication, which was clearly recommended by international and Chinese PD guidelines. But the PD depression treatment status in Chinese clinical practice is not systematically analyzed before. In this study, investigator will summarize the treatment profile of PD depression to see if PD depression is properly treated according to guideline.

ELIGIBILITY:
Inclusion Criteria:

* The incidence of depression in patients of Parkinson's disease (DSM-5 diagnostic criteria for depression)

Exclusion Criteria:

* Inability to understand or answer questions for any reason，that would interfere our assessment.
* Participate in a concurrent clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The estimated proportion of depression in patients with PD is around 50%. With 500 patients, the length of 95% CI of proportion of depression in PD patients will be less than 0.09 (the widest 95% confidence interval 0.088 will be attained only when the estimated proportion is 50%).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of depression in patients of Parkinson's disease (DSM-5 diagnostic criteria for depression) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Liu, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (4):
- China (4):
  - Department of Neurology,Nanjing Brain Hospital,Nanjing Medical University, Nanjing
  - Department of Neurology, Longhua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai
  - Department of Neurology, Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai
  - Zhongshan Hospital & Shanghai Medical College, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gan J, Zhou M, Chen W, Liu Z. Non-motor symptoms in Chinese Parkinson's disease patients. J Clin Neurosci. 2014 May;21(5):751-4. doi: 10.1016/j.jocn.2013.07.015. Epub 2013 Sep 11. PMID 24411328